CLINICAL TRIAL: NCT01907360
Title: A Phase I/II, Single Center, Single-Treatment, Open-Label, Adaptive Clinical Trial Design Examining the Pharmacokinetic Effects of up to Two Separate HLD200 Modified Release Formulations of Methylphenidate in Adolescent and Pediatric Subjects With ADHD
Brief Title: Pharmacokinetics of HLD200 in Children and Adolescents With ADHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ironshore Pharmaceuticals and Development, Inc (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLD200-102
Record Dates: First submitted 2013-07-12; First posted 2013-07-24 (Estimated); Results first posted 2021-09-20 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Attention-Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Intervention Model Description: Open-label, single-treatment
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HLD200 (methylphenidate hydrochloride) in Adolescents (Experimental): HLD200 (B formulation, 54 mg, oral capsules) administered as a single treatment in the evening to children aged 13-17 years.
  Interventions: Drug: HLD200 (methylphenidate hydrochloride)
- HLD200 (methylphenidate hydrochloride) in Children (Experimental): HLD200 (B formulation, 54 mg, oral capsules) administered as a single treatment in the evening to children aged 6-12 years.
  Interventions: Drug: HLD200 (methylphenidate hydrochloride)

INTERVENTIONS:
Drug: HLD200 (methylphenidate hydrochloride)
  Other Names: JORNAY PM

SUMMARY:
This study was designed to assess the pharmacokinetic effects of a single dose of HLD200 (methylphenidate hydrochloride) in children and adolescents with ADHD.

DETAILED DESCRIPTION:
This study utilized a single-center, open-label, single-treatment, fasted design to examine the rate and extent of absorption of evening-administered HLD200 in children (6-12 years) and adolescents (13-17 years) with ADHD.

Following a screening period that included five days washout to allow for clearance of any prior ADHD medications, subjects were domiciled in-clinic and administered HLD200 (B-formulation; 54 mg; oral capsule) at 9 pm under fasted conditions. Subjects were then observed for safety and tolerability and a total of 18 blood samples collected during a 48 hour period (at t=0, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24, 36 and 48 hours post-dosing). These samples were then assayed for methylphenidate plasma concentrations and this data used for calculation of pharmacokinetic parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents (13-17 years) and children (6-12 years).
* Previous diagnosis of ADHD and confirmation using the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
* ADHD symptoms controlled on a stable dose of ADHD medication. Subjects should be on MPH or have previous history of symptom control during treatment with MPH.
* Physical examination free of clinically significant findings, unless deemed NCS by the Investigator and Medical Monitor;
* Able to swallow treatment capsules;
* Available for entire study period;
* Provision of informed consent (from the parent[s] and/or legal representative[s]) and assent (from the subject); and
* Female subjects of childbearing potential (i.e., post-menarche) required to have a negative result on urine pregnancy testing (and will be given specific instructions on avoiding pregnancy during trial)

Exclusion Criteria:

* Any known history or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, ophthalmologic disease, unless deemed NCS by the Investigator and the Medical Monitor;
* Presence of any significant physical or organ abnormality;
* Any illness during the 4 weeks before this study, unless deemed NCS by the Investigator and the Clinical and/or Medical Monitor;
* Severe comorbid psychiatric diagnosis that may affect subject safety or confound results (e.g., psychosis, bipolar disorder);
* Known history of moderate to severe asthma;
* Known history of severe allergic reaction (including drugs, food, insect bites, environmental allergens);
* Known history of seizures (except febrile seizures prior to age 5), anorexia nervosa, bulimia or current diagnosis or family history of Tourette's disorder;
* Subject who are severely underweight or overweight.
* Clinical value outside of the acceptable ranges, unless deemed NCS significant per the Investigator;
* Positive history for hepatitis B, hepatitis C and Human Immunodeficiency Virus (HIV);
* Positive screening for illicit drug use, and/or current health conditions or use of medications that might confound the results of the study or increase risk to the subject;
* Use of prescription medications (except ADHD medications) within 7 days and over-the counter medications (except birth control) within the 3 days preceding study enrollment, unless deemed acceptable by the Investigator and Clinical and/or Medical Monitor;
* Blood draws of 50 ml to 249 ml within the 30 days, 250 ml to 449 ml within the 45 days and ≥ 450 ml within the 60 days preceding study enrollment;
* Participation in clinical trial with an investigational drug within the 30 days preceding study enrollment;
* Intolerance to venipuncture; and
* Current suicidal ideation or history of suicidality determined as a significant finding on the Columbia-Suicide Severity Rating Scale (C-SSRS) by the investigator (Baseline C-SSRS for adolescents; Pediatric Baseline C-SSRS for children).

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2013-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Childress, M.D., Principal Investigator — Centre for Psychiatry & Behavioral Medicine, Inc.
Locations (1):
- Centre for Psychiatry & Behavioral Medicine, Inc., Las Vegas, Nevada, United States

REFERENCES:
- [Derived] Childress A, Mehrotra S, Gobburu J, McLean A, DeSousa NJ, Incledon B. Single-Dose Pharmacokinetics of HLD200, a Delayed-Release and Extended-Release Methylphenidate Formulation, in Healthy Adults and in Adolescents and Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2018 Feb;28(1):10-18. doi: 10.1089/cap.2017.0044. Epub 2017 Oct 17. PMID 29039979

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 29 subjects were enrolled (18 adolescents and 11 children in sequential cohorts). Following consent/assent and screening procedures, subjects were required to wash-out of all ADHD medications for 5 days prior clinic admission for testing.
Groups:
- Adolescents (13-17yrs); Children (6-12 Yrs): Drug: B-HLD200 54mg capsules (Methylphenidate Modified Release B Formulation) or Drug: C-HLD200 54mg capsules (Methylphenidate Modified Release C Formulation)
  B-HLD200 54mg capsules
  C-HLD200 54mg capsules
Period: Overall Study
Arm/Group | Adolescents (13-17yrs) | Children (6-12 Yrs)
Started | 18 | 11
Completed | 18 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HLD200 (Methylphenidate Hydrochloride) in Adolescents: HLD200 (B formulation, 54 mg, oral capsules) administered as a single treatment in the evening to adolescents aged 13-17 years.
- Total: Total of all reporting groups
Arm/Group | HLD200 (Methylphenidate Hydrochloride) in Adolescents | HLD200 (Methylphenidate Hydrochloride) in Children | Total
Number analyzed (Participants) | 18 | 11 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.4 (1.24) | 10.5 (1.37) | 13.52 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 14 | 5 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 15 | 9 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 13 | 7 | 20
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 1 | 1 | 2
Height (cm) [Mean (Standard Deviation); unit: cm] | 169.56 (6.487) | 143.18 (6.072) | 159.55 (14.434)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 67.71 (14.588) | 36.08 (7.950) | 54.74 (19.704)

OUTCOME MEASURES:

1. Primary Outcome: PK Parameters for Rate and Extent of Absorption of MPH: Lag Time
Description: The absorption lag time for methylphenidate in plasma expressed in hours is the difference in time between the drug administration and the last time point where the drug concentration was below the limit of assay quantitation.
Time Frame: 48hrs
Population: All enrolled subjects included in analysis population.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- HLD200 in Adolescents (13-17 Years): Drug: HLD200 (methylphenidate hydrochloride; 54 mg) capsules
- HLD200 in Children (6-12 Yrs): Drug: HLD200 (methylphenidate hydrochloride; 54mg) capsules
Arm/Group | HLD200 in Adolescents (13-17 Years) | HLD200 in Children (6-12 Yrs)
Number analyzed (Participants) | 18 | 11
hours | 6.3 (1.3) | 3.3 (2.7)

2. Primary Outcome: PK Parameters for Rate and Extent of Absorption of MPH: Cmax
Description: The maximum drug concentration of methylphenidate in plasma.
Time Frame: 48hrs
Population: All enrolled subjects included in analysis population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | HLD200 in Adolescents (13-17 Years) | HLD200 in Children (6-12 Yrs)
Number analyzed (Participants) | 18 | 11
ng/mL | 7.17 (1.7) | 11.64 (4.2)

3. Primary Outcome: PK Parameters for Rate and Extent of Absorption of MPH: Tmax
Description: The time to reach maximum concentration of methylphenidate in plasma.
Time Frame: 48hrs
Population: All enrolled subjects included in analysis population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | HLD200 in Adolescents (13-17 Years) | HLD200 in Children (6-12 Yrs)
Number analyzed (Participants) | 18 | 11
hours | 17.1 (2.5) | 17.7 (2.5)

4. Primary Outcome: PK Parameters for Rate and Extent of Absorption of MPH: AUC0-tz
Description: Area under the methylphenidate plasma concentration-time curve to time point tz (AUC0-tz), where tz was the last time point over the time interval with a measurable drug concentration
Time Frame: 48hrs
Population: All enrolled subjects included in analysis population.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | HLD200 in Adolescents (13-17 Years) | HLD200 in Children (6-12 Yrs)
Number analyzed (Participants) | 18 | 11
ng.hr/mL | 105.5 (31.7) | 205.6 (80.4)

5. Primary Outcome: PK Parameters for Rate and Extent of Absorption of MPH: AUC0-inf
Description: The area under the methylphenidate plasma concentration-time curve to infinite time
Time Frame: 48hrs
Population: All enrolled subjects included in analysis population.
Measure: Mean (Standard Deviation); unit: ng.hr/mL
Arm/Group | HLD200 in Adolescents (13-17 Years) | HLD200 in Children (6-12 Yrs)
Number analyzed (Participants) | 18 | 11
ng.hr/mL | 109.6 (33.8) | 210.1 (80.9)

6. Other Pre Specified Outcome: PK Parameters for Rate and Extent of Absorption of MPH in Plasma: Plasma Concentration-time Curve
Description: To determine the rate and extent of absorption of methylphenidate following a single treatment of HLD200 (B formulation; 54 mg) in children and adolescents with ADHD, plasma samples were collected at t=0, 4, 6, 8, 9, 10, 11, 12, 13, 14, 15, 16, 18, 20, 22, 24, 36 and 48 hours post-HLD200 treatment and methylphenidate concentrations were determined.
Time Frame: 48hrs
Population: All enrolled subjects included in analysis population.
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | HLD200 in Adolescents (13-17 Years) | HLD200 in Children (6-12 Yrs)
Number analyzed (Participants) | 18 | 11
(ng/mL)
  t=0 hrs | 0.00 (0.00) | 0.00 (0.00)
  t=4 hrs | 0.00 (0.00) | 0.05 (0.07)
  t=6 hrs | 0.03 (0.06) | 0.13 (0.13)
  t=8 hrs | 0.15 (0.11) | 0.39 (0.21)
  t=9 hrs | 0.47 (0.36) | 1.03 (0.66)
  t=10 hrs | 1.37 (0.89) | 2.15 (1.41)
  t=11 hrs | 2.33 (1.32) | 4.42 (2.77)
  t=12 hrs | 3.76 (1.89) | 6.84 (4.01)
  t= 13 hrs | 4.66 (2.06) | 8.10 (4.72)
  t=14 hrs | 5.70 (2.02) | 9.05 (4.40)
  t=15 hrs | 6.09 (1.90) | 9.68 (4.06)
  t=16 hrs | 6.58 (1.57) | 10.64 (4.51)
  t=18 hrs | 6.13 (1.43) | 11.01 (3.90)
  t=20 hrs | 5.52 (1.56) | 10.53 (4.23)
  t=22 hrs | 4.66 (1.57) | 9.22 (3.76)
  t=24 hrs | 3.67 (1.70) | 7.51 (3.48)
  t=36 hrs | 1.07 (0.76) | 2.47 (1.05)
  t=48 hrs | 0.23 (0.30) | 0.48 (0.20)

ADVERSE EVENTS:
Time Frame: Baseline to 48 hours after the HLD200 dose
Groups:
- Adolescents (13-17yrs); Children (6-12 Yrs): Drug: B-HLD200 54mg capsules (Methylphenidate Modified Release B Formulation) or Drug: C-HLD200 54mg capsules (Methylphenidate Modified Release C Formulation)
Arm/Group | Adolescents (13-17yrs) | Children (6-12 Yrs)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/11
Other Adverse Events (participants affected / at risk) | 10/18 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adolescents (13-17yrs) (N=18) | Children (6-12 Yrs) (N=11)
Cerumen Impaction (Ear and labyrinth disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Musculoskeletal And Connective Tissue Disorders (Infections and infestations) | 1 | 0
Myalgia (Infections and infestations) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 2
Dizziness Postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No